CLINICAL TRIAL: NCT00522262
Title: Alberta Physical Activity and Breast Cancer Prevention (ALPHA) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other); University of Alberta (Other); University of Calgary (Other)
Responsible Party: Principal Investigator, Christine Friedenreich, Scientific Leader and Principal Investigator, AHS Cancer Control Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16649
Record Dates: First submitted 2007-08-27; First posted 2007-08-29 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Breast Neoplasms
Keywords: Breast Neoplasms; Exercise; Physical activity; Estrone; Estradiol; Adiposity; Breast density; Mammographic density; Insulin-Like Growth Factor I; Insulin Resistance; Women; Postmenopause
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Women randomized to the exercise intervention arm completed a one year aerobic exercise intervention of 225 minutes/week.
  Interventions: Behavioral: Aerobic exercise intervention
- Control (No Intervention): Women randomized to the control arm were asked to maintain their regular lifestyle which meant no changes to their exercise or dietary intake. Women eligible for this trial were inactive and hence were expected not to increase their levels of physical activity in the control arm.

INTERVENTIONS:
Behavioral: Aerobic exercise intervention — Women in the exercise arm underwent a year-long exercise intervention of five days per week of 45 minutes/session of moderate-vigorous intensity aerobic exercise.
  Arms: Exercise

SUMMARY:
The purpose of the ALPHA Trial is to examine the physiologic changes that occur in a woman's body when she begins exercising that may be related to a change in her risk of getting breast cancer.

DETAILED DESCRIPTION:
The goal of this study is to examine how a one-year exercise intervention, as compared to a usual sedentary lifestyle, influences specific biologic mechanisms that are hypothesized to be operative in the association between physical activity and breast cancer risk. These biologic mechanisms include sex hormone concentrations (estrone, estradiol and sex-hormone binding globulin); measures of adiposity and obesity; mammographic density; insulin-like growth factors; and insulin resistance.

A two-centered, two-armed randomized controlled trial (RCT) of exercise and risk factors for breast cancer will be conducted. Approximately 334 postmenopausal, sedentary women will be recruited to the study. Participants will be randomized to one of two groups: an exercise intervention, or a control group. The intervention group will undertake five weekly exercise sessions of 60 minutes each; three will be facility-based and two will be home-based each week. The Edmonton and Calgary exercise oncology facilities will be working in collaboration, and each will include both the controls and exercise intervention arms of the trial. The exercise intervention will last for 12 months. The control group will be asked not to change their usual level of activity during that time.

Baseline assessments will be obtained of serum sex hormones (estrone and estradiol), measures of obesity and adiposity, mammographic density, serum insulin growth factor (IGF)-1, insulin resistance, aerobic capacity, and psychosocial health measures. At the end of the study, all baseline assessments will be repeated and compared between the two groups.

This study will specifically address identified gaps in knowledge, in terms of examining the simultaneous effect of physical activity on several biologic mechanisms in a controlled trial setting, building on evidence from the only other randomized controlled trial on this topic. Strengths of the proposal include the multi-centered setting (utilizing facilities in both Calgary and Edmonton), and the collaboration of an experienced multi-disciplinary research team from across North America.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 50-74 at baseline
* Postmenopausal
* Moderately sedentary lifestyle
* Live in Calgary or Edmonton, Alberta, Canada
* English-speaking
* Willing to be randomized
* Body-mass index 22.0-40.0
* Breast tissue density >=0%

Exclusion Criteria:

* Previous invasive cancer in last 5 years
* Major co-morbidities
* Unable to participate in exercise program
* Current smoker
* Current excessive drinker
* Hormone replacement therapy use in previous 2 years
* Drugs that may influence one or more study outcomes

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 320 (Actual)
Dates: Start 2002-06; Primary Completion 2006-06 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Changes in estrone, estradiol and adiposity levels | Up to 12 months
  The effect of the exercise intervention on sex steroid and adiposity levels after one year is examined.

SECONDARY OUTCOMES:
Changes in mammographic density, insulin resistance and inflammatory markers | Up to 12 months
  The effect of the exercise intervention after one year is examined.
The effect of the exercise intervention on exercise adherence and quality of life. | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christine M Friedenreich, PhD, Principal Investigator — Alberta Health services
Locations (2):
- Canada (2):
  - Alberta Cancer Board, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

REFERENCES:
- [Result] Friedenreich CM, Woolcott CG, McTiernan A, Ballard-Barbash R, Brant RF, Stanczyk FZ, Terry T, Boyd NF, Yaffe MJ, Irwin ML, Jones CA, Yasui Y, Campbell KL, McNeely ML, Karvinen KH, Wang Q, Courneya KS. Alberta physical activity and breast cancer prevention trial: sex hormone changes in a year-long exercise intervention among postmenopausal women. J Clin Oncol. 2010 Mar 20;28(9):1458-66. doi: 10.1200/JCO.2009.24.9557. Epub 2010 Feb 16. PMID 20159820
- [Derived] Boyne DJ, King WD, Brenner DR, McIntyre JB, Courneya KS, Friedenreich CM. Aerobic exercise and DNA methylation in postmenopausal women: An ancillary analysis of the Alberta Physical Activity and Breast Cancer Prevention (ALPHA) Trial. PLoS One. 2018 Jun 28;13(6):e0198641. doi: 10.1371/journal.pone.0198641. eCollection 2018. PMID 29953441
- [Derived] McNeil J, Brenner DR, Courneya KS, Friedenreich CM. Dose-response effects of aerobic exercise on energy compensation in postmenopausal women: combined results from two randomized controlled trials. Int J Obes (Lond). 2017 Aug;41(8):1196-1202. doi: 10.1038/ijo.2017.87. Epub 2017 Mar 31. PMID 28360432
- [Derived] Friedenreich CM, Pialoux V, Wang Q, Shaw E, Brenner DR, Waltz X, Conroy SM, Johnson R, Woolcott CG, Poulin MJ, Courneya KS. Effects of exercise on markers of oxidative stress: an Ancillary analysis of the Alberta Physical Activity and Breast Cancer Prevention Trial. BMJ Open Sport Exerc Med. 2016 Oct 24;2(1):e000171. doi: 10.1136/bmjsem-2016-000171. eCollection 2016. PMID 27900199
- [Derived] Aparicio-Ting FE, Farris M, Courneya KS, Schiller A, Friedenreich CM. Predictors of physical activity at 12 month follow-up after a supervised exercise intervention in postmenopausal women. Int J Behav Nutr Phys Act. 2015 May 5;12:55. doi: 10.1186/s12966-015-0219-z. PMID 25940342
- [Derived] Woolcott CG, Courneya KS, Boyd NF, Yaffe MJ, McTiernan A, Brant R, Jones CA, Stanczyk FZ, Terry T, Cook LS, Wang Q, Friedenreich CM. Association between sex hormones, glucose homeostasis, adipokines, and inflammatory markers and mammographic density among postmenopausal women. Breast Cancer Res Treat. 2013 May;139(1):255-65. doi: 10.1007/s10549-013-2534-x. Epub 2013 Apr 21. PMID 23605145
- [Derived] Friedenreich CM, Neilson HK, Woolcott CG, Wang Q, Stanczyk FZ, McTiernan A, Jones CA, Irwin ML, Yasui Y, Courneya KS. Inflammatory marker changes in a yearlong randomized exercise intervention trial among postmenopausal women. Cancer Prev Res (Phila). 2012 Jan;5(1):98-108. doi: 10.1158/1940-6207.CAPR-11-0369. Epub 2011 Oct 7. PMID 21982875
- [Derived] Courneya KS, Tamburrini AL, Woolcott CG, McNeely ML, Karvinen KH, Campbell KL, McTiernan A, Friedenreich CM. The Alberta Physical Activity and Breast Cancer Prevention Trial: quality of life outcomes. Prev Med. 2011 Jan;52(1):26-32. doi: 10.1016/j.ypmed.2010.10.014. Epub 2010 Nov 8. PMID 21070806
- [Derived] Woolcott CG, Courneya KS, Boyd NF, Yaffe MJ, Terry T, McTiernan A, Brant R, Ballard-Barbash R, Irwin ML, Jones CA, Brar S, Campbell KL, McNeely ML, Karvinen KH, Friedenreich CM. Mammographic density change with 1 year of aerobic exercise among postmenopausal women: a randomized controlled trial. Cancer Epidemiol Biomarkers Prev. 2010 Apr;19(4):1112-21. doi: 10.1158/1055-9965.EPI-09-0801. Epub 2010 Mar 23. PMID 20332266